CLINICAL TRIAL: NCT00813059
Title: Intravitreal Bevacizumab for Treatment of the Second Eye With Non-Arteritic Ischemic Optic Neuropathy
Brief Title: Intravitreal Bevacizumab for Non-Arteritic Anterior Ischemic Optic Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Edward Margolin, MD, Mount Sinai Hospital, Canada
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: edmargolin
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Non-arteritic Anterior Ischemic Optic Neuropathy
Keywords: NAION; bevacizumab
MeSH Terms: conditions — Optic Neuropathy, Ischemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Intra-vitreal injection of bevacizumab (1.25mg/0.05ml)

INTERVENTIONS:
Drug: Intra-vitreal injection of bevacizumab (1.25mg/0.05ml) — Pars plana intra-vitreal injection of bevacizumab (1.25 mg/0.05 ml)

SUMMARY:
Non-Arteritic Ischemic Optic Neuropathy (NAION) is a disease producing swelling of the optic nerve (the "cable" going from the eye to the brain) resulting in decreased vision. About 15% of patients will experience NAION in the second eye; many of these patients will be left legally blind.

Currently, there is no treatment for NAION and for patients in whom the second eye becomes involved by the disease the outcome can be devastating.

The investigators are conducting a study where the investigators will inject a medication into the involved eye of patients with NAION. This medication might decrease the swelling of the optic nerve and improve their vision in that eye.

DETAILED DESCRIPTION:
NAION produces an ischemic insult in the optic nerve head presumably due to the hypoperfusion of the short ciliary arteries that supply it. This leads to the release of vascular endothelial growth factor (VEGF) and swelling of the affected area of the nerve. Vascular endothelial growth factor (VEGF) causes a rapid and reversible increase in vascular permeability and thus vasogenic edema of the affected area of the optic nerve head. Subsequently, increased pressure from the swelling of the affected segment causes compression and infarction of the previously not affected parts of the optic nerve by creating a sort-of "compartment syndrome".

Bevacizumab is a known anti-Vascular Endothelial Growth Factor (VEGF) agent. It is the investigators hypothesis that by injecting bevacizumab intra-vitreally the vasogenic edema will be reduced, preserving viable but threatened optic nerve tissue. One recent case report described a patient with sequential NAION treated with intra-vitreal bevacizumab who demonstrated significant improvement in visual acuity and on visual field testing (1). An editorial in the same issue of the Journal of Neuro-Ophthalmology in which this article appeared suggested that if the small studies evaluating intra-vitreal injections of bevacizumab in NAION would support its use in this disease, a large multi-center trial could be planned (2).

Intra-vitreal injections of bevacizumab have proven to be very safe in treatment of age-related macular degeneration (3). Because the patients that the investigators are planning to enroll in this study are faced with the real possibility of blindness with no therapeutic modality currently available to improve their visual outcome, the investigators believe that offering them intra-vitreal bevacizumab injection that might halt the progression of the visual acuity and visual field loss if our hypothesis is correct, would greatly improve their chances of avoiding blindness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed NAION (within the past 30 days but preferably within the first 14).

Exclusion Criteria:

* Patients who are unable to give informed consent
* Patient with:

  * uncontrolled glaucoma
  * pregnancy
  * lactation
  * proliferative diabetic retinopathy
  * active clinically significant diabetic macular edema
  * active uveitis
  * prior treatment with intraocular steroids that incited significant increase in intra-ocular pressure
  * other known causes of decreased visual acuity in the recently involved eye such as significant dry or wet macular degeneration
  * previous history of other optic neuropathies
  * previous history of ocular trauma that resulted in decreased visual acuity
* Patients with baseline amblyopia in the newly involved eye and visual acuity worse than 20/50 prior to the onset of NAION
* Previous treatment for any ocular condition with any investigational drugs

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who gained three or more lines of vision at six months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Margolin, Principal Investigator — Mount Sinai Hospital, University of Toronto
Locations (1):
- Mount Sinai Hospital, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bennett JL, Thomas S, Olson JL, Mandava N. Treatment of nonarteritic anterior ischemic optic neuropathy with intravitreal bevacizumab. J Neuroophthalmol. 2007 Sep;27(3):238-40. doi: 10.1097/WNO.0b013e31814b273d. No abstract available. PMID 17895825
- [Background] Kelman SE. Intravitreal triamcinolone or bevacizumab for nonarteritic anterior ischemic optic neuropathy: do they merit further study? J Neuroophthalmol. 2007 Sep;27(3):161-3. doi: 10.1097/WNO.0b013e31814a61ae. No abstract available. PMID 17895813
- [Background] Fung AE, Rosenfeld PJ, Reichel E. The International Intravitreal Bevacizumab Safety Survey: using the internet to assess drug safety worldwide. Br J Ophthalmol. 2006 Nov;90(11):1344-9. doi: 10.1136/bjo.2006.099598. Epub 2006 Jul 19. PMID 16854824